CLINICAL TRIAL: NCT02449070
Title: Effects of Nicorandil on Cardiac Infarct Size in Patients With ST-segment Elevation Acute Myocardial Infarction : A Randomized Clinical Trial
Brief Title: Effects of Nicorandil on Cardiac Infarct Size in Patients With ST-segment Elevation Acute Myocardial Infarction
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pusan National University Hospital (Other)
Collaborators: JW Pharmaceutical (Industry)
Responsible Party: Principal Investigator, Jun-Hyok OH, Assistant professor, Pusan National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D-1407-011-030
Record Dates: First submitted 2015-05-13; First posted 2015-05-20 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Myocardial Infarction
Keywords: Nicorandil; Cardiac MRI
MeSH Terms: conditions — Myocardial Infarction | interventions — Nicorandil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nicorandil (Experimental): Receive nicorandil before primary PCI and thereafter for 6 months along with the standard therapy.
  Interventions: Drug: Nicorandil
- Control (No Intervention): Receive primary PCI and the standard therapy.

INTERVENTIONS:
Drug: Nicorandil — 4 mg iv after randomization, 2 mg ic just before ballooning, 2 mg ic just before stenting
  Other Names: Nicrodandil
  Arms: Nicorandil

SUMMARY:
The purpose of this study is to determine whether nicorandil reduce cardiac infarct size in patient with ST-segment elevation acute myocardial infarction.

DETAILED DESCRIPTION:
Study objective :

To investiage whether nicorandil treatment reduce infarct size measured by cardiac MRI at 6 months after primary PCI

Allocation :

1. Nicorandil arm :

   Recieve nicorandil 4 mg i.v. before undergoing PCI, additionall 2mg i.c. just before 1st ballooning, additionall 2mg i.c. just before stenting, After successful PCI, 10 mg/day (or 5 mg/day) p.o. for 6 months.
2. Control arm :

Recieve standard treatment including PCI, but avoid nicoranil and adenosine.

Follow-up and Measurement :

Cardiac MRI scans are scheduled at 5 days and 6 months after primary PCI. Clinically followed upto 6 months after parimary PCI.

ELIGIBILITY:
Inclusion Criteria:

* STEMI patients presenting within 12 hours after symptom onset
* Undergoing primary PCI

Exclusion Criteria:

* Previous myocardial infarction
* Atrial fibrillation
* RV infarction
* Cardiogenic shock
* Serum creatinine >2.0 mg/dL
* Narrow angle glaucoma
* Taking PDE-5 inhibitors

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2015-05; Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Infarct size as measured by cardiac MRI | Six months after primary PCI

SECONDARY OUTCOMES:
LVEF(%) as measured by cardiac MRI | Five days and 6 months after primary PCI
MVO as measured by cardiac MRI | Five days after primary PCI
ST-segment resolution | One hour after primary PCI
MACE (Death, Spontaneous MI, Stroke) | up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jun-Hyok Oh, MD, Principal Investigator — Pusan National University Hospital
Locations (1):
- Pusan National University Hospital, Pusan, South Korea